CLINICAL TRIAL: NCT05596825
Title: Phenotypic Characteristics of Responders to Obstructive Sleep Apnea Treatment Using Mandibular Advancement Devices
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: sacagon
Record Dates: First submitted 2022-10-10; First posted 2022-10-27 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2022-10

CONDITIONS: Sleep Apnea
Keywords: sleep apnea syndrome; mandibular advancement device
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Occlusal Splints

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Mandibular Advancement Device — To analyze the phenotypic characteristics of different subgroups of patients with obstructive sleep apnea syndrome who respond better (complete responders) or worse (partial responders or non-responders) to treatment with mandibular advancement devices.
  Responders will be defined as a post-treatment AHI of less than 10/h and at least a 50 percent reduction in their AHI. Partial responders will be defined as a post-treatment AHI greater than 10/hour but at least a 50 percent reduction in AHI, and non-responders as less than a 50 percent reduction compared to baseline.

SUMMARY:
Currently, mandibular advancement devices (MAD) are recommended by the American Academy of Sleep Medicine (AASM) as the first treatment a line in cases of mild and moderate OSAS in patients without severe cardiovascular comorbidity and in severe OSAS when treatment with CPAP fails or is rejected. Although oral appliances (OD) have less impact on AHI reduction, both treatments have been shown to have a similar impact on clinical outcomes, including symptomatology and cardiovascular outcomes. In addition, MAD is a treatment that is better tolerated by patients, which results in greater compliance on their part, and therefore a similar efficacy in clinical practice.

Its mechanism of action consists of maintaining the patency of the upper airway, preventing collapse. They act by correcting the anatomical imbalance of patients with OSAS, specifically stabilizing and increasing the space of the velopharyngeal airways, reducing their collapsibility.

However, the effectiveness of the treatment of this pathology using MAD is limited by the inter-individual preference of the results of the treatment and the lack of information in the correct selection of the appropriate patients. In fact, oral appliances are an effective treatment for 60-70% of patients. Therefore, the precise selection of patients is essential to optimize the results of MAD treatment and thus avoid the necessary costs. This justifies the need to identify phenotypes likely to predict response to MAD treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Adult patients with obstructive sleep apnea diagnosed according to the third edition of the International Classification of Sleep Disorders.
* Apnea-hypopnea index (AHI) of at least 5/hour of sleep.

Exclusion Criteria:

* Patients with heart disease.
* Central sleep apnea.
* Patients who had degenerative pathologies of the temporomandibular joint.
* Patients who had moderate or advanced periodontal disease.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Master's Degree in Prosthodontics and Occlusion at the University of Valencia will be selected. At the dental clinic of the Lluis Alcanyis Foundation. Located in Gascó Oliag Nº 1, Valencia.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-07-08 (Estimated); Primary Completion 2023-12-08 (Estimated); Study Completion 2024-04-29 (Estimated)

PRIMARY OUTCOMES:
Gender | 1 day
  Male or Female
Age | 1 day
  Age described as "years and months". The age of the patients at the beginning of the study
Body mass index | 1 day
  Weight and height will be combined to report BMI in kg/m^2. The body mass index at the beginning of the study.
Epworth Daytime Sleepiness Scale | 1 day
  The ESS is a self-administered questionnaire that evaluates sub- jective daytime sleepiness in quotidian situations. The score ranges from 0 to 24 and is usually elevated in sleep apnea patients, indicating a propensity to fall asleep. An ESS score above 10 is considered abnormal and a maximum score of 24 indicates severe somnolence.
Anatomical characteristics | 12 months
  Craniofacial and airway features from cone beam computed tomography. (eg. maxillary length (mm), mandibular length (mm), anterior facial height (mm), posterior facial height (mm), distance between hyoid bone and mandibular plane (mm), distance between retrognation point and mandibular plane (mm), upper airway length (mm), superior airway space (mm) and inferior airway space (mm)).
apnea - hypopnea index | 6 months
  number of apnea and hypopnea per hours of sleep before and after the device's placement.
minimum oxygen saturation | 6 months
  It is the minimum oxyhemoglobin saturation during a sleep study. Expressed in %.

IPD SHARING:
Plan to Share IPD: No